CLINICAL TRIAL: NCT01599390
Title: Burden of Influenza in the United States, July 1997 up to April 2009
Brief Title: Influenza Burden Assessment in the United States, July1997 - up to April 2009
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Sage Analytica (Industry)
Responsible Party: Sponsor
Other Study IDs: 116730
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Influenza
Keywords: United States; Burden of Disease; Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Data Collection

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Influenza Group
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — The study will use multiple primary data sources: the Nationwide Inpatient Sample (for hospitalisations) and the US National Vital Statistics System (for mortality), and weekly virology data from the Centers for Disease Control and Prevention (CDC) influenza surveillance program supplemented with literature data.
  Weekly time series of the rates of various severe influenza-related health outcomes will be constructed. Statistical models, guided by weekly numbers of cases of laboratory-confirmed influenza and respiratory syncytial virus (RSV) contained in the CDC virology data, will be constructed to estimate the portions of the various outcomes that can be attributed to influenza. Next, the seasonal impact of influenza by age, risk status, and influenza subtype will be assessed. Finally, the potential burden that a quadrivalent vaccine could have prevented over the 12 year study period will be predicted.

SUMMARY:
The study will assess the burden of severe influenza outcomes by age, risk status, and influenza subtype, in order to create a profile of the burden of influenza-related morbidity and mortality in United States from July 1997 to April 2009.

DETAILED DESCRIPTION:
This epidemiological study is a modelling of time series retrospectively extracted from multiple databases. Data will be extracted from existing electronic healthcare databases.

ELIGIBILITY:
Inclusion Criteria:

* Recorded in the US NIS hospitalization data or the US National Vital Statistics System (NVSS) mortality data with a pre-specified diagnostic code.

Exclusion Criteria:

* Missing data in the following fields: age, primary discharge diagnosis, admission month (NIS) /month of death (NVSS), and status at discharge (alive / dead).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All records of people in the US in the Nationwide Inpatient Sample (NIS) hospitalization data or in the US mortality data will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Occurrences of potentially influenza-attributable hospitalization or death by age, risk status, region and season. | From July 1997 to April 2009 (i.e., up to almost 12 years)
Amount of circulating influenza A and B, and RSV strains determined for each season. | From July 1997 to April 2009 (i.e., up to almost 12 years)

SECONDARY OUTCOMES:
Influenza vaccine content and effectiveness by season. | From July 1997 to April 2009 (i.e., up to almost 12 years)
Influenza vaccine coverage by season. | From July 1997 to April 2009 (i.e., up to almost 12 years)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Matias G, Taylor R, Haguinet F, Schuck-Paim C, Lustig R, Shinde V. Estimates of hospitalization attributable to influenza and RSV in the US during 1997-2009, by age and risk status. BMC Public Health. 2017 Mar 21;17(1):271. doi: 10.1186/s12889-017-4177-z. PMID 28320361